CLINICAL TRIAL: NCT07116889
Title: A Phase 1 First in Human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of GB-0895 in Adults With Mild to Moderate Asthma or Single Dose in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Investigate GB-0895 in Adults With Mild to Moderate Asthma or COPD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Generate Biomedicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GB-0895-101; 2023-507611-35-00 (EU CTIS Number); 1008606 (Registry Identifier: Integrated Research Application System (IRAS))
Record Dates: First submitted 2025-07-23; First posted 2025-08-12 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Asthma; COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Generate Biomedicines
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Ascending Dose (SAD) (asthma participants) (Experimental): randomized 3:1 active:placebo
  Interventions: Biological: GB-0895 (SC); Drug: Placebo (SC)
- Part B: Multiple Ascending Dose (MAD) (asthma participants) (Experimental): randomized 3:1 active:placebo
  Interventions: Biological: GB-0895 (SC); Drug: Placebo (SC)
- Part C: Single Dose (COPD participants) (Experimental): randomized 3:1 active:placebo
  Interventions: Biological: GB-0895 (SC); Drug: Placebo (SC)

INTERVENTIONS:
Biological: GB-0895 (SC) — Single subcutaneous dose of GB-0895
  Arms: Part A: Single Ascending Dose (SAD) (asthma participants); Part C: Single Dose (COPD participants)
Biological: GB-0895 (SC) — Multiple subcutaneous doses of GB-0895
  Arms: Part B: Multiple Ascending Dose (MAD) (asthma participants)
Drug: Placebo (SC) — Single subcutaneous dose of placebo
  Arms: Part A: Single Ascending Dose (SAD) (asthma participants); Part C: Single Dose (COPD participants)
Drug: Placebo (SC) — Multiple subcutaneous doses of placebo
  Arms: Part B: Multiple Ascending Dose (MAD) (asthma participants)

SUMMARY:
This study is testing the safety, tolerability, pharmacokinetics and pharmacodynamics of GB-0895.

ELIGIBILITY:
Inclusion Criteria (Part A & B, Asthma):

* Participants must be able to give written consent
* 18 to 65 years of age (inclusive) at the screening visit;
* Diagnoses of mild to moderate asthma for ≥12 months
* Laboratory blood values within the ranges outlined in the protocol

Exclusion Criteria (Part A & B, Asthma):

* Other serious disease
* Significant asthma exacerbations
* Current smokers or ex-smokers with >5 pack years smoking history
* Pregnant or breastfeeding

Inclusion Criteria (Part C, COPD):

* Participants must be able to give written consent
* 40 to 80 years of age (inclusive) at the screening visit;
* Diagnoses of COPD for ≥12 months
* Laboratory blood values within the ranges outlined in the protocol
* Must be current or ex-smoker

Exclusion Criteria (Part C, COPD):

* Other serious disease
* COPD exacerbation within 4 weeks of enrolling
* Requires supplemental oxygen (CPAP for sleep apnea allowed)
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE 5.0 | Day 1 to Day 500

SECONDARY OUTCOMES:
Measure of maximum plasma concentration of GB-0895 | Day 1 to Day 500
Total exposure of GB-0895 (AUC) | Day 1 to Day 500
Blood eosinophil counts | Day 1 to Day 500
Incidence of treatment-emergent anti-drug antibody (ADA) response | Day 1 to Day 500

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - Alcanza, DeLand, Florida
  - Miami Research Institute of South Florida, Miami, Florida
  - Omega Research, Orlando, Florida
  - Nucleus Network, Saint Paul, Minnesota
  - Southeastern Research Center, Winston-Salem, North Carolina
  - DM Clinical Research, Tomball, Texas
- Germany (3):
  - Charite Research Organization GmbH, Berlin
  - IKF Pneumologie, Frankfurt
  - Fraunhofer Institut fur Toxikologie and Experimentelle Medizin (ITEM), Hanover
- United Kingdom (4):
  - Hammersmith Medicines Research, London
  - Queen Anne Street Medical Center, London
  - Medicines Evaluation Unit (MEU), Manchester
  - Simbec-Orion Clinical Development, Merthyr Tydfil

IPD SHARING:
Plan to Share IPD: No